CLINICAL TRIAL: NCT03741036
Title: Immediate Implant Placement With Provisionalization Using Autogenous Bone Graft Particulates vs Deproteinized Bovine Bone vs Nano-hydroxyapatite Alloplast as a Space Filling Material in the Maxillary Esthetic Zone
Brief Title: Immediate Implant Placement With Provisionalization Using Different Bone Grafts as a Space Filling Material in the Maxillary Esthetic Zone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mohamed tarek mohamed youssif omar (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Mohamed tarek mohamed youssif omar, Researcher, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-27-7-2018
Record Dates: First submitted 2018-10-19; First posted 2018-11-14 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Dental Implant Failed
Keywords: immidiate; dental implant; immidiate provisionalization; bone graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- autogenous bone graft as a space filling material (Active Comparator): Autogenous bone from sub mental bone had been grafted in jumping gap between implant and freshely extracted socket
  Interventions: Procedure: Autogenous bone graft as space filling in immidiate implant placment
- deproteinized bovine as a space filling material (Active Comparator): Granules of deproteinized bovine bone of 0.25-1.0 mm diameter were used to fill the remaining defect when the distance of the defect wall to the implant surface was > 3 mm.
  Interventions: Procedure: Deprotinized bovien as space filling in immidate implant placement
- nano-hydroxyapatite alloplast as a space filling material (Active Comparator): The patient was treated using alloplast material mixed with a nano-bone graft to fill gap between implant and freshely extracted socket
  Interventions: Procedure: Nano-hydroxiapatite alloplast in immidiate implant placement

INTERVENTIONS:
Procedure: Autogenous bone graft as space filling in immidiate implant placment — * The selected patients will be informed of the nature of the research work and informed consent will be obtained (immediate implant placement grafting with autogenous bone graft)
  * Patients will be subjected to CBCT (diagnostic for upper arch).
  * Local anesthesia will be given to the patient.
  * Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
  * The procedure will be carried out flapless.
  * In the study group: Atraumatic extraction
  * The extraction socket will be evaluated for absence of any fenestration or granulation tissues
  Arms: autogenous bone graft as a space filling material
Procedure: Deprotinized bovien as space filling in immidate implant placement — * The selected patients will be informed of the nature of the research work and informed consent will be obtained (immediate implant placement grafting with deprotinized bovien material)
  * Patients will be subjected to CBCT (diagnostic for upper arch).
  * Local anesthesia will be given to the patient.
  * Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
  * The procedure will be carried out flapless.
  * In the study group: Atraumatic extraction
  * The extraction socket will be evaluated for absence of any fenestration or granulation tissues
  Arms: deproteinized bovine as a space filling material
Procedure: Nano-hydroxiapatite alloplast in immidiate implant placement — * The selected patients will be informed of the nature of the research work and informed consent will be obtained (immediate implant placement grafting with nano-hydroxiapatite alloplast material )
  * Patients will be subjected to CBCT (diagnostic for upper arch).
  * Local anesthesia will be given to the patient.
  * Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
  * The procedure will be carried out flapless.
  * In the study group: Atraumatic extraction
  * The extraction socket will be evaluated for absence of any fenestration or granulation tissues
  Arms: nano-hydroxyapatite alloplast as a space filling material

SUMMARY:
compare autogenous bone graft, xenograft and nanohydroxyapatite in immediate implant w placement in maxillary esthetic zone with provisionalization

DETAILED DESCRIPTION:
Placement of implants into extraction sockets targets the maintenance of peri implant hard and soft tissue structures and the support of a natural and esthetic contour. The main advantages of immediate implant insertion in comparison with delayed implant placement protocols are as follows: a reduced treatment time, less number of sessions, and, thus, the less invasive procedure. This study examines the clinical performance (survival rate, marginal bone levels and Pink Esthetic Score [PES]) of OsseoSpeed™ implants placed into extraction sockets with immediate provisionalization in the anterior maxilla after a follow-up of at least 12 months.

The removal of teeth results inevitably in both horizontal and vertical changes of hard and soft tissue dimensions.

Clinical research has shown that the loss of volume in the extraction sockets is high: the biggest bone volumetric changes take place during the first 12 months from the dental extraction, with a reduction of bone volume of 50%, of which 2/3 (30%) are within the first 3 months.

Nowadays to get success in postextraction implantology means managing the early and irreversible alveolar bone dimensional changes following tooth extraction, in order to minimize the negative effects on the aesthetics final.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with badly broken teeth in upper esthetic zone indicated for extraction
* Both sexes.
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placemen

Exclusion Criteria:

* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems
* Disorders to implant are related to history of radiation therapy to the head and neck neoplasia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-27 (Estimated); Primary Completion 2019-07-27 (Estimated); Study Completion 2019-08-17 (Estimated)

PRIMARY OUTCOMES:
Primary stability (marginal bone loss) | 3 months
  measure device (osstell )

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University, Cairo
  - Mohamed tarek, Cairo

IPD SHARING:
Plan to Share IPD: Undecided